CLINICAL TRIAL: NCT04175912
Title: A Phase 2 Study of Pevonedistat in Combination With Carboplatin and Paclitaxel in Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Testing the Combination of Pevonedistat With Chemotherapy for Bile Duct Cancer of the Liver
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-07769; NCI-2019-07769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2187 (Other: ECOG-ACRIN Cancer Research Group); EA2187 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Cholangiocarcinoma; Metastatic Hepatocellular Carcinoma; Stage III Hepatocellular Carcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIA Hepatocellular Carcinoma AJCC v8; Stage IIIA Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIB Hepatocellular Carcinoma AJCC v8; Stage IIIB Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Hepatocellular Carcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Stage IVA Hepatocellular Carcinoma AJCC v8; Stage IVB Hepatocellular Carcinoma AJCC v8; Unresectable Cholangiocarcinoma; Unresectable Hepatocellular Carcinoma; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular | interventions — Carboplatin; Paclitaxel; Taxes; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (pevonedistat) (Experimental): Patients receive pevonedistat IV over 60 minutes on days 1, 3, and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pevonedistat
- Arm B (pevonedistat, paclitaxel, carboplatin) (Experimental): Patients receive pevonedistat IV over 1 hour on days 1, 3, and 5, paclitaxel IV over 3 hours on day 1, and carboplatin IV over 15-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Starting cycle 5, patients may receive pevonedistat monotherapy at the discretion of treating physician.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pevonedistat

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm B (pevonedistat, paclitaxel, carboplatin)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (pevonedistat, paclitaxel, carboplatin)
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924

SUMMARY:
This phase II trial studies how well pevonedistat alone or in combination with chemotherapy (paclitaxel and carboplatin) works in treating patients with bile duct cancer of the liver. Pevonedistat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This study may help the study doctors find out how well pevonedistat shrinks bile duct cancer of the liver when given alone and when in combination with paclitaxel and carboplatin.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate of pevonedistat as a single agent and in combination with carboplatin and paclitaxel in patients with unresectable intrahepatic cholangiocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of pevonedistat alone and in combination with carboplatin and paclitaxel in patients with intrahepatic cholangiocarcinoma.

II. To determine the clinical benefit rate of patients with advanced intrahepatic cholangiocarcinoma (ICC) treated with pevonedistat monotherapy and in combination with carboplatin and paclitaxel.

III. To determine progression-free survival of patients treated with pevonedistat monotherapy and in combination with carboplatin and paclitaxel.

IV. To determine overall survival of patients treated with pevonedistat monotherapy and in combination with carboplatin and paclitaxel.

EXPLORATORY OBJECTIVES:

I. To determine whether overexpression of NEDD8, NAE1, and UBC12 predict response to treatment.

II. To identify the mutation profile of those cholangiocarcinomas with overexpression of the neddylation pathway.

III. To bank specimens for further future investigations.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive pevonedistat intravenously (IV) over 60 minutes on days 1, 3, and 5. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive pevonedistat IV over 1 hour on days 1, 3, and 5, paclitaxel IV over 3 hours on day 1, and carboplatin IV over 15-60 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Starting cycle 5, patients may receive pevonedistat monotherapy at the discretion of treating physician.

After completion of study treatment, patients are followed up at 30 days after last dose of study treatment, then every 3 months for the first year and every 6 months for years 2-3.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patient must have a life expectancy >= 12 weeks
* Patient must have histologically confirmed intrahepatic cholangiocarcinoma or biphasic hepatocellular carcinoma and cholangiocarcinoma that is metastatic or unresectable and who have progressed on or been intolerant of one prior line of systemic gemcitabine containing chemotherapy regimen.

  * NOTE: Prior immunotherapy or targeted therapies are allowed and will not be considered a line of therapy unless administered with cytotoxic chemotherapy
* Patient must have measurable disease. For patients who have received localized therapy (embolization, chemoembolization, radiofrequency ablation or radiation) are eligible if measurable disease is not within the treatment field or the treated disease has clearly progressed since last localized therapy
* Leukocytes >= 3,000/mcL (obtained within 14 days prior to randomization)
* Absolute neutrophil count >= 1,500/mcL (obtained within 14 days prior to randomization)
* Platelets >= 100,000/mcL (obtained within 14 days prior to randomization)
* Total bilirubin =< institutional upper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may enroll if direct bilirubin =< 1.5 x ULN of the direct bilirubin (obtained within 14 days prior to randomization)
* Hemoglobin >= 9 g/dL (obtained within 14 days prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained within 14 days prior to randomization)
* Creatinine =< institutional ULN, OR glomerular filtration rate (GFR) >= 40 mL/min/1.73 m^2 (obtained within 14 days prior to randomization)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Known HIV positive patients who meet the following criteria will be considered eligible:

  * CD4 count >= 350 cells/mm^3
  * Undetectable viral load
  * Maintained on modern therapeutic regimens utilizing non-CYP interactive agents (i.e. excluding ritonavir)
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients who received prior platinum or taxane chemotherapy are eligible
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. In addition, patients with any of the known cardiopulmonary disease, defined as follows, would be ineligible for this trial:

  * Unstable angina
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV;);
  * Myocardial infarction within 6 months prior to randomization (patients who had ischemic heart disease such as acute coronary syndrome [ACS], myocardial infarction, and/or revascularization greater than 6 months before randomization and who are without cardiac symptoms may enroll)
  * Symptomatic cardiomyopathy
  * Clinically symptomatic pulmonary hypertension requiring pharmacologic therapy
  * Clinically significant arrhythmia, defined as:

    * History of polymorphic ventricular fibrillation or torsade de pointes,
    * Permanent atrial fibrillation, defined as continuous atrial fibrillation for >= 6 months,
    * Persistent atrial fibrillation, defined as sustained atrial fibrillation lasting > 7 days and/or requiring cardioversion in the 4 weeks before randomization,
    * Grade 3 atrial fibrillation defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation
    * Patients with paroxysmal atrial fibrillation or grade < 3 atrial fibrillation for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Participants with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible

Exclusion Criteria:

* Patients must not have had major surgery within 14 days before randomization. Patients with surgery planned during study period are ineligible
* Women must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. Patients must also not expect to conceive or father children from the time of registration, while on study treatment, and until at least 4 months after the last dose of study treatment. All females of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential and sexually active males must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and continue for at least 4 months after the last dose of protocol treatment
* Male patients must not donate sperm during the course of this study or within 4 months after receiving their last dose of protocol treatment
* Female patients must not donate eggs (ova) during the course of this study or within 4 months after receiving their last dose of protocol treatment
* Patient must not have a prolonged rate corrected QT (QTc) interval >= 480 msec calculated according to institutional guideline
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e. have residual toxicities > grade 1) are ineligible with the exception of alopecia
* Patients with persistent >= grade 2 diarrhea lasting more than 3 days within 14 weeks of randomization are ineligible
* Patients with known central nervous system (CNS) involvement are ineligible
* Patients must not be receiving any other investigational agents
* Patients must not have received chemotherapy or radiotherapy within 2 weeks prior to randomization. Prior treatment with radiation therapy involving >= 25% of hematopoietically active bone marrow will be ineligible
* Patients must not have received immunotherapy within 8 weeks prior to randomization
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to pevonedistat, carboplatin, or paclitaxel
* Patient must not be receiving any treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of the study drug as below. Clinically significant metabolic enzyme inducers are not permitted during the study. Patients must not be receiving any medications or substances that are strong inducers of CYP3A4/5 (i.e. phenytoin, rifampin, St. Johns wort) or inhibitors of breast cancer resistance protein (BCRP) (i.e. cyclosporine). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if a new medication need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Inhibitors of CYP3A4/5 are allowed
* Patients must not have uncontrolled intercurrent illness
* Patients must not have uncontrolled coagulopathy or bleeding disorder
* Patients must not have active, uncontrolled infection or severe infectious disease such as severe pneumonia, meningitis, or septicemia
* Patients with known moderate chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis are ineligible
* Patients must not have psychiatric illness/social situations that would limit compliance with study requirements
* Participants must not have had prior pevonedistat treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2026-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Deming, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (421):
- United States (421):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Mercy Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Holy Name Hospital, Teaneck, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of North Carolina-Hillsborough Campus, Hillsborough, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 patients were enrolled between March 16, 2020 and March 22, 2023.
Period: Overall Study
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
Started | 20 | 20
Received Treatment | 17 | 17
Eligible and Treated | 17 | 17
Completed | 0 | 0
Not Completed | 20 | 20
Not completed — Disease progression- relapse during active treatment | 17 | 13
Not completed — Adverse Event | 0 | 3
Not completed — Never started treatment | 3 | 3
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Median (Full Range); unit: years] | 63.4 [43.7 to 73.7] | 62.3 [34.0 to 78.9] | 63.1 [34.0 to 78.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 10 | 15 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: Response was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Objective response includes complete response (CR) and partial response (PR).
  CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 3 months for the first year and every 6 months for years 2-3
Population: Eligible and treated patients are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 17 | 17
Participants
  With Objective Response | 0 | 0
  Without Objective Response | 17 | 17

2. Secondary Outcome: Clinical Benefit
Description: Clinical benefit was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1), including complete response (CR), partial response (PR) and stable disease (SD) that lasted greater than or equal to 24 weeks.
  CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Every 3 months for the first year and every 6 months for years 2-3
Population: Eligible and treated patients are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 17 | 17
Participants
  With Clinical Benefit | 0 | 1
  Without Clinical Benefit | 17 | 16

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to progression or death, whichever came first; patients alive without evidence of disease progression were censored at the date of last disease assessment. Patients who died without documented progression and the death occurred > 6 weeks of last disease assessment will be censored at the date of last disease assessment that showed progression-free.
  Progression was evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1), defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions is also considered as progression.
Time Frame: Every 3 months for the first year and every 6 months for years 2-3
Population: Eligible and treated patients are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 17 | 17
months | 1.54 [1.41 to 2.10] | 2.92 [1.71 to 5.55]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause, and patients still living were censored at the date last known alive.
Time Frame: Every 3 months for the first year and every 6 months for years 2-3
Population: Eligible and treated patients are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 17 | 17
months | 4.80 [4.04 to 12.50] | 6.54 [4.20 to 14.80]

5. Other Pre Specified Outcome: Associations Between Response and Overexpression of NEDD8, NAE1, and UBC12
Description: Associations between response and overexpression of NEDD8, NAE1, and UBC12 will be evaluated.
Time Frame: Assessed every 3 months for the first year and every 6 months for years 2-3
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Mutation Profile of Those Cholangiocarcinomas
Description: To identify the mutation profile of those cholangiocarcinomas with overexpression of the neddylation pathway
Time Frame: Assessed at baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Specimens Banking
Description: To bank specimens for further future investigations
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Incidence of Adverse Event
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment, up to 3 years
Description: All treated patients are included in this analysis.
Arm/Group | Arm A (Pevonedistat) | Arm B (Pevonedistat, Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 17/17 | 15/17
Serious Adverse Events (participants affected / at risk) | 8/17 | 12/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Pevonedistat) (N=17) | Arm B (Pevonedistat, Paclitaxel, Carboplatin) (N=17)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Death NOS (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 0 | 2
Disease progression (General disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Hepatic infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
INR increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Pevonedistat) (N=17) | Arm B (Pevonedistat, Paclitaxel, Carboplatin) (N=17)
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 7 | 11
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 3
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Edema limbs (General disorders) | 1 | 5
Fatigue (General disorders) | 14 | 17
Fever (General disorders) | 3 | 3
Flu like symptoms (General disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 2 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 8
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 8
Ascites (Gastrointestinal disorders) | 3 | 0
Bloating (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 6 | 9
Diarrhea (Gastrointestinal disorders) | 2 | 8
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 6 | 11
Stomach pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Hepatic infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Herpes simplex reactivation (Infections and infestations) | 1 | 0
Thrush (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 13
Alkaline phosphatase increased (Investigations) | 5 | 7
Aspartate aminotransferase increased (Investigations) | 6 | 12
Blood bilirubin increased (Investigations) | 5 | 4
Cardiac troponin I increased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 0 | 1
Creatinine increased (Investigations) | 2 | 4
GGT increased (Investigations) | 5 | 6
INR increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 7 | 7
Neutrophil count decreased (Investigations) | 1 | 6
Platelet count decreased (Investigations) | 3 | 11
Weight loss (Investigations) | 3 | 0
White blood cell decreased (Investigations) | 2 | 10
Blood bicarbonate decreased (Investigations) | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 8 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 7 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 4
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 4 | 2
Paresthesia (Nervous system disorders) | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 12
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 4 | 6
Depression (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 3 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Urine discoloration (Renal and urinary disorders) | 2 | 0
Glucosuria (Renal and urinary disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 3
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 5 | 5
Thromboembolic event (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04175912/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04175912/ICF_001.pdf